CLINICAL TRIAL: NCT07293819
Title: Comprehensive Assessment of First Trimester Pregnancy Loss: Analyzing Its Impact and Biological Pathways to Develop Tailored Management Care Strategies (The FIRST-CARE Study)
Brief Title: Comprehensive Assessment of First Trimester Pregnancy Loss
Acronym: FIRST-CARE
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Cristina Trilla, MD, PhD - Consultant in Obstetrics and Gynecology, Clinical Coordinator of the Pregnancy Loss Functional Unit, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-FIR-2024-199; PI24/01735 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2025-07-20; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Miscarriage in First Trimester
Keywords: Miscarriage; First-trimester; Genetic testing; angiogenic markers; pregnancy loss; perinatal grief; reproductive immunology; anti-phospholipid syndrom; cell-free DNA; chorionic villous sampling
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Chorionic villous sampling, blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: First Miscarriage Cohort: Women who have experienced their first clinically confirmed first-trimester miscarriage (n=150).
- Group 2: Recurrent Pregnancy Loss (RPL) Cohort: Women with a history of two or more first-trimester miscarriages (n=75).

SUMMARY:
The FIRST-CARE Study is a prospective research project conducted at Hospital de la Santa Creu i Sant Pau (Barcelona, Spain), aimed at better understanding the causes and consequences of first-trimester pregnancy loss (miscarriage).

Miscarriage is a common event that affects about 15% of clinically recognized pregnancies and can have both physical and emotional consequences for women and their partners. However, many questions about its causes remain unanswered, and most women do not receive a clear explanation or personalized support after experiencing a loss.

This study will include 225 women who have experienced a miscarriage during the first 14 weeks of pregnancy. Two groups will be studied: those who have had a miscarriage for the first time and those with a history of recurrent pregnancy loss (defined as two or more previous miscarriages). The aim is to investigate a wide range of possible causes - including genetic, hormonal, immune, cardiovascular, placental, and psychological factors - in order to improve diagnosis and develop more personalized care strategies.

Participants will undergo a comprehensive evaluation including ultrasound, blood tests, genetic testing, and psychological assessments. In some cases, their partners will also be invited to participate. Women will be followed for one year to assess their mental well-being and reproductive outcomes, such as the chance of getting pregnant again and the outcome of future pregnancies.

The study will also create a biobank of biological samples to support future research in the field of pregnancy loss.

By combining clinical evaluations, laboratory tests, and personal experiences, this study aims to uncover new insights into why miscarriages happen and how to better support women and couples going through this experience. The ultimate goal is to provide better diagnostic tools, care pathways, and support systems to reduce the emotional burden of miscarriage and improve reproductive health outcomes.

DETAILED DESCRIPTION:
Background and Rationale Miscarriage, or early pregnancy loss, is the most common complication of pregnancy, affecting approximately 15% of clinically recognized gestations. However, this percentage is likely underestimated, as many early losses occur before the pregnancy is even detected by ultrasound. Miscarriage is often considered a sporadic event, but in many cases it can be the first sign of underlying health issues that affect maternal, paternal, or embryonic health.

Despite its frequency, miscarriage remains poorly understood and inconsistently investigated. Women experiencing early pregnancy loss often receive no clear explanation, no thorough assessment, and no tailored follow-up or support. In recurrent cases (recurrent pregnancy loss, RPL), the diagnostic work-up is limited and typically reserved for women who have had at least two or three losses. This approach leaves many women without answers and without the opportunity to benefit from early intervention or support.

Miscarriage also carries significant emotional and psychological consequences, which are often underestimated. Research has shown associations between miscarriage and depression, anxiety, post-traumatic stress, and even long-term health risks, including cardiovascular disease. Addressing miscarriage as both a biological and psychosocial condition is critical to improving patient care and outcomes.

Study Aim

The FIRST-CARE Study (First Trimester Comprehensive Assessment and Reproductive Evaluation) is a prospective, single-center cohort study designed to investigate the biological, clinical, and psychological dimensions of first-trimester miscarriage. The study aims to:

1. Identify preventable or treatable causes of early pregnancy loss.
2. Characterize maternal and paternal health factors involved in miscarriage.
3. Understand the emotional impact and mental health consequences of miscarriage.
4. Develop tailored diagnostic and management strategies based on biological pathways and patient needs.

Study Population

The study will enroll 225 women with a diagnosis of first-trimester missed miscarriage (up to 14 weeks gestation), divided into two groups:

* Group A: 150 women experiencing their first miscarriage.
* Group B: 75 women with a history of recurrent pregnancy loss (≥2 miscarriages).

Exclusion criteria include multiple pregnancy, ectopic pregnancy, and molar pregnancy. Male partners will also be invited to participate in selected assessments.

Study Procedures

Participants will undergo a comprehensive evaluation consisting of the following components:

1. Genetic Testing of Pregnancy Loss

   Chorionic villus sampling (CVS) for karyotyping, microarray, and QF-PCR of products of conception.

   Fetal cell-free DNA analysis from maternal blood to assess chromosomal abnormalities in cases where CVS is not feasible.

   Evaluation of test performance and genetic diagnostic yield by gestational age and recurrence status.
2. Maternal Health Assessment

   Detailed obstetric and gynecological history.

   Gynecological ultrasound (2D/3D) and uterine artery Doppler.

   Measurement of angiogenic markers (PlGF, sFlt-1) and cardiovascular indicators (NT-proBNP).

   Endocrinological testing: thyroid function, insulin resistance, glucose metabolism, Vitamin D levels, progesterone.

   Immunological testing: antiphospholipid antibodies, thyroid antibodies, ANA, lymphocyte populations, KIR/HLA compatibility, GDF-15.
3. Paternal Evaluation

   Age, BMI, medical comorbidities, lifestyle factors (smoking, alcohol, diet, exercise).

   Semen analysis.
4. Psychological and Social Assessment

Evaluation of depressive symptoms (EPDS), grief (Perinatal Grief Scale), PTSD (PCL-5), quality of life (SF-36), coping strategies (COPE-28), and social support (MSPSS).

Assessment of stigma, self-compassion, and experiential avoidance. Qualitative interviews conducted by a psychologist and midwife to understand the lived experience of miscarriage and care needs.

Biological Sample Collection

* Maternal and paternal blood, chorionic villi, urine, vaginal and rectal swabs for future research.
* All samples will be stored in a biobank following participant consent.

Follow-Up and Outcomes

Participants will be followed up for one year to evaluate:

Psychological recovery and well-being. Subsequent reproductive outcomes, including new pregnancies and their outcomes (e.g., preeclampsia, fetal growth restriction, preterm birth).

Comparative prevalence of biological factors in first vs. recurrent loss.

Follow-up visits include:

Psychological assessment at 1 month and 1 year post-loss. Clinical and laboratory assessments at 6-12 weeks post-loss. Data on future pregnancies will be collected throughout the year following enrollment.

Expected Results and Impact

The FIRST-CARE Study is designed to fill several critical gaps in the current understanding and management of early pregnancy loss:

* From the First Loss: By including women at the first miscarriage, the study will explore whether biological differences exist between first and recurrent losses and assess whether earlier interventions could reduce recurrence and long-term morbidity.
* Comprehensive Assessment: The study goes beyond standard protocols by incorporating advanced genetic, immunological, and placental markers, many of which are not routinely evaluated in clinical practice.
* Biological Pathways: Investigating the interactions between maternal, paternal, and placental factors will help elucidate the underlying pathophysiology of miscarriage and support the development of individualized diagnostic and therapeutic approaches.
* Psychological and Social Support: Assessing mental health and psychosocial stressors will inform the design of better counseling strategies and highlight the importance of emotional support in miscarriage care.

Ethics and Confidentiality The study has been approved by the Ethics Committee of Hospital de la Santa Creu i Sant Pau. All participants will provide written informed consent. Data will be coded, stored securely, and handled according to the General Data Protection Regulation (EU 2016/679) and Spanish data protection laws. Only anonymized data will be used in scientific publications and presentations.

The procedures involved in the study are considered low-risk and are either standard of care or non-invasive. Chorionic villus sampling will be offered only after appropriate counseling and consent. Participants will be offered the option to receive their results, and their clinical care will not be altered by study participation.

Data Analysis and Statistical Approach Data will be analyzed using descriptive and inferential statistics. Multivariate models will be developed to identify predictive factors for miscarriage and assess the relationship between clinical variables and outcomes. In addition, advanced statistical techniques such as Bayesian Kernel Machine Regression (BKMR) will be used to explore complex interactions among biological variables.

Dissemination and Future Perspectives The findings of the FIRST-CARE Study will be published in peer-reviewed journals and presented at international conferences in reproductive medicine and women's health. A biobank of samples will be created to support future investigations. The study will also contribute to national and international clinical guidelines on the evaluation and care of early pregnancy loss.

Ultimately, this research aims to change the clinical approach to miscarriage, promote earlier and more compassionate care, reduce recurrence, and empower women and couples with knowledge and support during one of the most challenging experiences in reproductive life.

ELIGIBILITY:
Female participants:

Inclusion Criteria:

* Women aged 18 years or older.
* Diagnosis of missed miscarriage in the first trimester (<14 weeks of gestation) confirmed by ultrasound.
* Presence of an intrauterine pregnancy with fetal demise (clinical pregnancy loss).
* Willing and able to provide written informed consent.
* Ability to understand and complete study procedures.

Exclusion Criteria:

* Multiple pregnancy (twins or more).
* Ectopic pregnancy.
* Molar pregnancy (complete or partial hydatidiform mole).
* Ongoing pregnancy with fetal cardiac activity.
* Inability or unwillingness to comply with study procedures or follow-up.

Male participants: no specific inclusion or exclusion criteria will apply to male partners, since the main inclusion criteria is a clinical pregnancy loss.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years or older with a diagnosis of first-trimester missed miscarriage (gestational age <14 weeks) will be enrolled. The study population will include two cohorts: women experiencing their first miscarriage and women with a history of recurrent pregnancy loss (defined as two or more previous first-trimester miscarriages). Participants will be recruited at the Hospital de la Santa Creu i Sant Pau (Barcelona, Spain) from outpatient and emergency gynecology services. Male partners will be invited to participate in selected assessments when applicable.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Composite Prevalence Index of Biological Risk Factors in First-Trimester Pregnancy Loss | Baseline to 3 months post-miscarriage
  Proportion of women with at least one biological abnormality among the following categories:
  1. Genetic (e.g., pathogenic or likely pathogenic variants identified by chromosomal microarray analysis or targeted gene panels),
  2. Immunologic (e.g., positive antiphospholipid antibodies, abnormal NK cell activity, ANA positivity),
  3. Endocrine (e.g., abnormal TSH, HOMA index, HbA1c or fasting glucose levels),
  4. Angiogenic or Cardiovascular (e.g., altered uterine artery Doppler indices, abnormal serum PlGF or sFlt-1).
  Abnormality is defined according to established clinical cutoffs for each parameter. The outcome is calculated as the percentage of participants with at least one abnormal result in any of the assessed categories.
  Comparison will be made between women with a first miscarriage and women with recurrent pregnancy loss (RPL).

SECONDARY OUTCOMES:
Prevalence of Genetic Abnormalities in Women with First-Trimester Pregnancy Loss | Baseline to 3 months post-miscarriage
  Evaluation of the proportion of women with pathogenic or likely pathogenic variants identified by chromosomal cytogenetics (karyotyping), microarray analysis (CMA) or cfDNA in the first miscarriage group versus the recurrent pregnancy loss group.
  Units of Measure: Percentage of participants (%)
Prevalence of Immunological Abnormalities in Women with First-Trimester Pregnancy Loss | Within 12 weeks after diagnosis of pregnancy loss
  Evaluation of the proportion of women with abnormal immunological markers (e.g., antiphospholipid antibodies, antibuclears antibodies (ANA), peripheral lymphocyte activity) using standardized immunoassays.
  Unit of measurement: positivity for ANA, NK cells > 12%, positivity for anti-phospholipid syndrom
Prevalence of of Endocrine Abnormalities | Within 12 weeks after diagnosis of pregnancy loss
  Proportion of women with abnormal thyroid function tests (TSH, T4), and/or abnormal glucose metabolism (HbA1c), and/or HOMA index.
  Unit measurements: TSH > 4mUI/L; HbA1c < 5.7%; HOMA index > 2.5
Frequency of Angiogenic and Cardiovascular Dysfunction | Within 12 weeks after diagnosis of pregnancy loss
  Presence of altered uterine artery Doppler indices > 2.5 or abnormal levels of angiogenic markers (e.g., PlGF, sFlt-1), measured by Doppler ultrasound and immunoassays.
Subsequent pregnancy rate and outcomes within 12 months | Up to 12 months after enrollment or until delivery of subsequent pregnancy
  Proportion of participants who achieve a new pregnancy and corresponding obstetric outcomes: miscarriage, preeclampsia, fetal growth restriction, gestational diabetes, preterm birth
Diagnostic yield of genetic testing (cfDNA vs. CVS) by gestational age and recurrence | At time of diagnosis
  Assessment of performance (informative vs. non-informative results) and concordance of genetic testing modalities in miscarriage diagnosis
Development of multivariate models for individual miscarriage risk stratification | After data completion (12 months)
  Use of multivariate and machine-learning models to identify predictive factors for miscarriage based on biological and clinical data
Depression Symptoms at 1 Month and 12 Months Post-Miscarriage | 1 month and 12 months after pregnancy loss
  Depression symptoms will be assessed using the Edinburgh Postnatal Depression Scale (EPDS).
  The EPDS is a 10-item self-report scale designed to screen for postnatal depression.
  Score range: 0-30, where higher scores indicate worse depressive symptoms. Scores ≥13 suggest probable depression. Unit of Measure: EPDS total score
Anxiety and Post-Traumatic Stress Symptoms at 1 Month and 12 Months Post-Miscarriage | 1 month and 12 months after pregnancy loss
  Post-traumatic stress symptoms will be assessed using the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5).
  The PCL-5 is a 20-item self-report measure of PTSD symptoms. Score range: 0-80, where higher scores indicate greater PTSD symptom severity. A cut-off score of 33 is commonly used for PTSD screening. Unit of Measure: PCL-5 total score
Grief Symptoms at 1 Month and 12 Months Post-Miscarriage | 1 month and 12 months after pregnancy loss
  Grief will be assessed using the Perinatal Grief Scale (PGS) - Short Form. This 33-item self-report questionnaire evaluates grief reactions specific to perinatal loss.
  Score range: 33-165, where higher scores reflect more intense grief. Unit of Measure: PGS-SF total score
Health-Related Quality of Life at 1 Month and 12 Months Post-Miscarriage | 1 month and 12 months after pregnancy loss
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36).
  The SF-36 provides eight domain scores and two summary scores (Physical and Mental Component Summary).
  Score range per domain: 0-100, where higher scores indicate better health status.
  Unit of Measure: SF-36 domain scores

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures may be shared with qualified researchers upon reasonable request and with appropriate data use agreements. Shared data may include clinical, laboratory, and questionnaire data, excluding any personal identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD), along with supporting documentation such as the study protocol, statistical analysis plan (SAP), and informed consent form (ICF), will be made available to qualified researchers upon reasonable request. Data will be shared after publication of the main study results and upon execution of a data use agreement.
  Data will be shared through institutional repositories or secure transfer methods in accordance with data protection regulations.
Access Criteria: Qualified researchers affiliated with academic institutions, hospitals, or public health organizations will be eligible to request access to de-identified individual participant data (IPD) and supporting documentation, including the study protocol, statistical analysis plan (SAP), and informed consent form (ICF).
  Access will be granted for scientifically sound research proposals that are compatible with the original study objectives or explore related topics in reproductive health and early pregnancy loss.
  Interested researchers must submit a data access request to the study sponsor or principal investigator. Upon approval, data will be shared under the terms of a data use agreement, which will outline responsibilities regarding data confidentiality, use, and publication.
  Data will be provided in electronic format via secure transfer platforms managed by the sponsor institution.